CLINICAL TRIAL: NCT05557006
Title: Change of QRS Morphology and Electrophysiological Characteristics During Pacing Within the Interventricular Septum: a Prospective, Observational Study
Brief Title: Change of QRS Morphology and Electrophysiological Characteristics During Pacing Within the Interventricular Septum
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Yanchun Liang, Prof., General Hospital of Shenyang Military Region
Other Study IDs: GHNTC-PACE
Record Dates: First submitted 2022-09-19; First posted 2022-09-27 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Cardiac Pacing
Keywords: Left Bundle Branch Pacing; Left Bundle Branch Area Pacing; Septal Pacing; Left Ventricular Activation Time; Right Ventricular Activation Time

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All patients: Patients who meet the inclusion criteria
  Interventions: Procedure: left bundle branch pacing

INTERVENTIONS:
Procedure: left bundle branch pacing — In the procedure of left bundle branch pacing, various QRS morphologies are observed as penetrating the lead into the interventricular septum.

SUMMARY:
Conduction system pacing (CSP), including His bundle pacing (HBP) and left bundle branch (LBB) pacing (LBBP), as a physiological pacing strategy, can achieve interventricular and/or intra-left ventricular mechanical synchronization by delivering physiological or nearly physiological ventricular activation. And many studies have verifed clinical efficacy of CSP that it can significantly relieve dyssynchrony of ventricular contraction, improve cardiac function and reduce the risk of heart failure as compared to right ventricular pacing. However, CSP has some shortcomings which limit its widespread application to some extent. As for HBP, although it can achieve optimal physiological ventricular synchronization, the problems of relatively high pacing threshold, low R-wave amplitude, the long-term performance, and inability to correct infra-Hisian atrioventricular block and intraventricular block in some patients have always been concerns. Nevertheless, LBBP is likely free of the restrictions mentioned above. On the contrary, LBBP can capture the left conduction system by directly stimulating the proximal LBB distal to the site of conduction block, thereby achieving rapid and physiological LV activation with a lower and stable pacing threshold and higher R-wave amplitude. However, as a newly emerged physiologic pacing technology, LBBP is currently in the exploratory stage and there are some phenomena to be interpreted, such as the evolution of pacing QRS morphology during the lead penetration into the interventricular septum. Therefore, the aim of this study is to assess the morphological evolution and electrophysiological characteristics of various pacing QRS patterns observed as the lead penetrates the interventricular septum from right to left.

ELIGIBILITY:
Inclusion Criteria:

* The indications for pacemaker implantation are in accordance with the 2021 European Society of Cardiology (ESC) guidelines.
* Patients requiring a high percentage of ventricular pacing (>40% expected ventricular pacing) include patients with advanced or third-degree atrioventricular block and atrial fibrillation with bradycardia.
* Left bundle branch pacing will be performed.
* Patients voluntarily participate and sign informed consent.

Exclusion Criteria:

* Atrioventricular block caused by reversible factors such as acute myocardial infarction and electrolyte disturbance.
* Patients with severe liver or renal failure.
* Life expectancy < 1 year.
* Patients with age < 18 years.
* Left ventricular ejection fraction (LVEF) < 40%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring a high percentage of ventricular pacing (>40% expected ventricular pacing) include patients with advanced or third-degree atrioventricular block and atrial fibrillation with bradycardia.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-09-27 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Left ventricular activation time (LVAT) | Continuous uninterrupted monitoring during the lead penetration into the interventricular septum.
  Left ventricular activation time (LVAT) is defined as the interval from the onset of the pacing stimulus to the peak of the R wave in lead V5/6, which reflects the lateral precordial myocardium depolarization time.
Right ventricular activation time (RVAT) | Continuous uninterrupted monitoring during the lead penetration into the interventricular septum.
  Right ventricular activation time (RVAT) is defined as the interval from the onset of the pacing stimulus to the peak potential recorded by the atrial electrode temporarily placed in the right ventricle, which reflects delayed right ventricular activation.
Paced QRS morphology | Continuous uninterrupted monitoring during the lead penetration into the interventricular septum.
  Paced QRS morphology during lead penetration through the interventricular septum mainly includes left bundle branch block, intraventricular block and right bundle branch block.

SECONDARY OUTCOMES:
Stimulus-QRSend duration (s-QRSend) | Continuous uninterrupted monitoring during the lead penetration into the interventricular septum.
  Stimulus-QRSend duration (s-QRSend) is the time from the onset of the pacing stimulus to the end of QRS complex.
The late-R wave duration and amplitude in lead V1 (r´dur、r´amp) | Continuous uninterrupted monitoring during the lead penetration into the interventricular septum.
  The late-R wave duration in lead V1 indicates delayed right ventricular excitation.
The S wave duration and amplitude in lead V6 (Sdur、Samp) | Continuous uninterrupted monitoring during the lead penetration into the interventricular septum.
  The S wave duration in lead V6 indicates delayed right ventricular excitation.

CONTACTS AND LOCATIONS:
Overall Officials: Yanchun Liang, MD、PhD, Principal Investigator — The General Hospital of Northern Theater Command
Locations (1):
- General Hospital of Northern Theater Command, Shenyang, Liaoning, China

REFERENCES:
- [Background] Shimeno K, Tamura S, Nakatsuji K, Hayashi Y, Abe Y, Naruko T. Characteristics and proposed mechanisms of QRS morphology observed during the left bundle branch pacing procedure. Pacing Clin Electrophysiol. 2021 Dec;44(12):1987-1994. doi: 10.1111/pace.14382. Epub 2021 Oct 31. PMID 34662435
- [Background] Zhang J, Sheng X, Pan Y, Wang M, Fu G. Electrophysiological Insights into Three Modalities of Left Bundle Branch Area Pacing in Patients Indicated for Pacing Therapy. Int Heart J. 2021 Jan 30;62(1):78-86. doi: 10.1536/ihj.20-490. Epub 2020 Dec 26. PMID 33390564